CLINICAL TRIAL: NCT03026322
Title: Preventing Hypoxemia With Manual Ventilation During Endotracheal Intubation (PreVent) Trial
Acronym: PreVent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Semler, Assistant Professor, Division of Pulmonary and Critical Care Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB #161962
Record Dates: First submitted 2017-01-16; First posted 2017-01-20 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Respiratory Failure; Respiratory Failure With Hypoxia; Endotracheal Intubation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — N(6)-2-(4-aminophenyl)ethyladenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Ventilation (Active Comparator): Beginning after the administration of sedation/neuromuscular blockade, manual ventilation will be provided by bag-valve-mask until the initiation of laryngoscopy. In patients requiring more than one attempt at laryngoscopy, bag-valve-mask ventilation will resume between laryngoscopy attempts.
  Interventions: Other: Manual Ventilation
- No Manual Ventilation (Active Comparator): Between the administration of sedation/neuromuscular blockade and intubation, ventilation will not be provided unless the patient experiences an arterial oxygen saturation less than 90%. For patients who experience an oxygen saturation less than 90% after induction, bag-valve-mask ventilation may be provided.
  Interventions: Other: No Manual Ventilation

INTERVENTIONS:
Other: Manual Ventilation — Beginning after the administration of sedation/neuromuscular blockade, manual ventilation will be provided by bag-valve-mask until the initiation of laryngoscopy. In patients requiring more than one attempt at laryngoscopy, bag-valve-mask ventilation will resume between laryngoscopy attempts.
  Other Names: Bag-valve-mask ventilation
  Arms: Manual Ventilation
Other: No Manual Ventilation — Between the administration of sedation/neuromuscular blockade and intubation, ventilation will not be provided unless the patient experiences an arterial oxygen saturation less than 90%. For patients who experience an oxygen saturation less than 90% after induction, bag-valve-mask ventilation may be provided.
  Other Names: Apnea
  Arms: No Manual Ventilation

SUMMARY:
Complications are common during endotracheal intubation of critically ill adults. Manual ventilation between induction and intubation ("bag-valve-mask" ventilation) has been proposed as a means of preventing hypoxemia, the most common complication of intubation outside the operating room. Safety and efficacy data, however, are lacking. PreVent is a randomized trial comparing manual ventilation between induction and laryngoscopy to no manual ventilation between induction an laryngoscopy during endotracheal intubation of critically ill adults. The primary efficacy endpoint will be the lowest arterial oxygen saturation. The primary safety endpoints will be the lowest oxygen saturation, highest fraction of inspired oxygen, and highest positive end-expiratory pressure in the 24 hours after the procedure.

DETAILED DESCRIPTION:
PreVent is a prospective, parallel-group, pragmatic, randomized trial comparing manual ventilation between induction and laryngoscopy to no manual ventilation between induction an laryngoscopy during endotracheal intubation of critically ill adults. The primary aim of the PreVent trial is to compare the effect of manual ventilation between induction and intubation versus no manual ventilation on the lowest arterial oxygen saturation experienced by critically ill adults undergoing endotracheal intubation. The PreVent trial is anticipated to begin enrollment in January 2017 and will enroll adults undergoing endotracheal intubation with sedation and/or neuromuscular blockade in participating units. Patients will be randomized 1:1 to manual ventilation versus no manual ventilation. In the manual ventilation group, manual ventilation using a bag-valve-mask will be provided from the time of induction until the time of endotracheal intubation, except during laryngoscopy. In the no manual ventilation group, no manual ventilation will be provided between induction and endotracheal intubation, except for the treatment of hypoxemia. The primary efficacy endpoint will be the lowest arterial oxygen saturation during the procedure. The primary safety endpoints will be the lowest oxygen saturation, highest fraction of inspired oxygen, and highest positive end expiratory pressure in the 24 hours after intubation. Conduct of the trial will be overseen by a Data Safety Monitoring Board. An interim analysis will be performed after the enrollment of 175 patients. The analysis of the trial will be conducted in accordance with a pre-specified statistical analysis plan made publicly available prior to the conclusion of enrollment. The initial planned enrollment of 350 patients was increased by the Data and Safety Monitoring Board at the interim analysis to a final planned enrollment of 400 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is located in a participating unit
* Planned procedure is endotracheal intubation
* Planned operator is a provider expected to routinely perform endotracheal intubation in the participating unit
* Administration of sedation and/or neuromuscular blockade is planned
* Age ≥ 18 years old

Exclusion Criteria:

* Urgency of intubation precludes safe performance of study procedures
* Operator feels a specific approach to ventilation between induction and intubation is required
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-05-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Lowest arterial oxygen saturation | Induction to 2 minutes after completion of the airway management procedure
  The lowest arterial oxygen saturation measured by continuous pulse oximetry (SpO2) between induction and 2 minutes after completion of the airway management procedure.

SECONDARY OUTCOMES:
Incidence of lowest oxygen saturation less than 90% | Induction to 2 minutes after completion of the airway management procedure
  Incidence of lowest oxygen saturation less than 90% in the time from induction to 2 minutes after completion of the airway management procedure.
Incidence of lowest oxygen saturation less than 80% | Induction to 2 minutes after completion of the airway management procedure
  Incidence of lowest oxygen saturation less than 80% in the time from induction to 2 minutes after completion of the airway management procedure.
Change in saturation from induction to lowest oxygen saturation | Induction to 2 minutes after completion of the airway management procedure
  Change in saturation from induction to lowest oxygen saturation within 2 minutes after completion of the airway management procedure.
Incidence of desaturation | Induction to 2 minutes after completion of the airway management procedure
  Incidence of desaturation as defined by a decrease in oxygen saturation of greater than 3% from induction to lowest oxygen saturation within 2 minutes after completion of the airway management procedure.
Lowest oxygen saturation in the 24 hours after intubation. | 24 hours after intubation
Highest fraction of inspired oxygen in the 24 hours after intubation. | 24 hours after intubation
Highest positive end expiratory pressure in the 24 hours after intubation. | 24 hours after intubation
Lowest oxygen saturation, highest fraction of inspired oxygen, and highest positive end expiratory pressure from 0-1, 1-6, and 6- 24 hours after intubation. | 24 hours after intubation
  Lowest oxygen saturation, highest fraction of inspired oxygen, and highest positive end expiratory pressure from 0-1, 1-6, and 6- 24 hours after intubation.
Operator-reported pulmonary aspiration | Induction to 2 minutes after completion of the airway management procedure
  Visualization of oropharyngeal or gastric contents in the pharynx, larynx, or trachea between induction and completion of airway management.
New infiltrate on chest imaging in the 48 hours after intubation | 48 hours after intubation
  Determination of new infiltrate will be made by two blinded experts (pulmonary/critical care attendings or fellows) with adjudication by a third expert in the case of discordant results
Operator-reported pulmonary aspiration, new chest x-ray infiltrate, OR lowest oxygen saturation < 80% (composite outcome) | 48 hours after intubation
New pneumothorax or pneumomediastinum on chest imaging in the 24 hours after intubation | 24 hours after intubation
Incidence of esophageal intubation | Induction to 2 minutes after completion of the airway management procedure
Lowest systolic blood pressure (peri-procedural) | Induction to 2 minutes after completion of the airway management procedure
  Lowest systolic blood pressure between induction and two minutes after completion of the airway management procedure
New systolic blood pressure < 65 mmHg or new need for vasopressor | Induction to 2 minutes after completion of the airway management procedure
  New systolic blood pressure < 65 mmHg or new need for vasopressor between medication administration and 2 minutes following successful placement of an endotracheal tube
Cardiac arrest within one hour of intubation | One hour after intubation.
Death within one hour of intubation | One hour after intubation
Cormack-Lehane grade of glottic view | Induction to 2 minutes after completion of the airway management procedure
Operator-assessed difficulty of intubation | Induction to 2 minutes after completion of the airway management procedure
Incidence of successful intubation on the first laryngoscopy attempt | Induction to 2 minutes after completion of the airway management procedure
Number of laryngoscopy attempts | Induction to 2 minutes after completion of the airway management procedure
Time from induction to successful intubation | Induction to 2 minutes after completion of the airway management procedure
Need for additional airway equipment or a second operator | Induction to 2 minutes after completion of the airway management procedure
In-hospital mortality | 28 days
Ventilator-free days | 28 days
  Ventilator-free days to day 28 will be defined as the number of days alive and with unassisted breathing to day 28 after enrollment, assuming a patient survives for at least two consecutive calendar days after initiating unassisted breathing and remains free of assisted breathing. If a patient returns to assisted breathing and subsequently achieves unassisted breathing prior to day 28, VFD will be counted from the end of the last period of assisted breathing to day 28. If the patient is receiving assisted ventilation at day 28 or dies prior to day 28, VFD will be 0. If a patient is discharged while receiving assisted ventilation, VFD will be 0. All data will be censored at the first of hospital discharge or 28 days.
Intensive care unit-free days | 28 days
  ICU-free days to 28 days after enrollment will be defined as the number of days alive and not admitted to an intensive care unit service after the patient's final discharge from the intensive care unit in that hospitalization before 28 days. Patients who are never discharged from the intensive care unit will receive a value of 0. Patients who die before day 28 will receive a value of 0. For patients who return to an ICU and are subsequently discharged prior to day 28, ICU-free days will be counted from the date of final ICU discharge. All data will be censored at the first of hospital discharge or 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Semler, MD, MSc, Study Director — Vanderbilt University Medical Center; Todd W Rice, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (5):
- United States (5):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Harborview Medical Center, University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Casey JD, Janz DR, Russell DW, Vonderhaar DJ, Joffe AM, Dischert KM, Brown RM, Zouk AN, Gulati S, Heideman BE, Lester MG, Toporek AH, Bentov I, Self WH, Rice TW, Semler MW; PreVent Investigators and the Pragmatic Critical Care Research Group. Bag-Mask Ventilation during Tracheal Intubation of Critically Ill Adults. N Engl J Med. 2019 Feb 28;380(9):811-821. doi: 10.1056/NEJMoa1812405. Epub 2019 Feb 18. PMID 30779528
- [Derived] Casey JD, Janz DR, Russell DW, Vonderhaar DJ, Joffe AM, Dischert KM, Brown RM, Lester MG, Zouk AN, Gulati S, Stigler WS, Rice TW, Semler MW; PreVent Investigators and the Pragmatic Critical Care Research Group. Manual ventilation to prevent hypoxaemia during endotracheal intubation of critically ill adults: protocol and statistical analysis plan for a multicentre randomised trial. BMJ Open. 2018 Aug 10;8(8):e022139. doi: 10.1136/bmjopen-2018-022139. PMID 30099400